CLINICAL TRIAL: NCT02926755
Title: Multi-modality Imaging in Acute Myocardial Infarction
Acronym: MIAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Robert Safian, MD., Corewell Health East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-144
Record Dates: First submitted 2016-08-15; First posted 2016-10-06 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Acute Myocardial Infarction; STEMI; Coronary Artery Disease; Atherosclerotic Plaque Disruption With Thrombosis of Artery
Keywords: Intra Venous Ultrasound (IVUS); Fractional Flow Reserve (FFR); Optical Coherence Tomography (OCT); Acute Myocardial Infarction; Coronary Artery Disease (CAD); Angiography
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Angiography to Assess Vulnerable Plaque (Experimental): In order to characterize plaque a repeat Coronary Angiography within 2 to 40 days will be done to assess vulnerable plaque features such as plaque tears, plaque thickness, plaque volume, and lipid content in plaque) in heart arteries in patients who have suffered a recent acute heart attack, and who have blockages >50% in one or more of the other arteries in the heart.
  Interventions: Procedure: Coronary Angiography

INTERVENTIONS:
Procedure: Coronary Angiography — Coronary angiography which includes fractional flow reserve (FFR),that allows precise measurement of blood flow in the arteries to the heart; the Near Infra-Red Spectroscopy-Intravascular Ultrasound (NIRS IVUS) provides information about the amount of lipid and cholesterol in the plaque, and plaque volume;the Optical Coherence Tomography (OCT) allows physicians to assess tears in the surface of plaque and plaque thickness; and Coronary CT Angiography (CCTA) to evaluate plaque characteristics, and correlate with the invasive findings. The research portion of the study requires all imaging studies be performed (NIRS, IVUS, OCT, FFR) during coronary angiography, rather than just one or two of these imaging studies, and the CCTA.

SUMMARY:
The goal of this study is to use three (3) different imaging techniques:Fractional Flow Reserve (FFR) allows precise measurement of blood flow in the arteries to the heart, and is more reliable than pictures alone to determine the significance of blockages in the heart; Near Infra-Red Spectroscopy-Intravascular Ultrasound (NIRS IVUS) provides information about the amount of lipid and cholesterol in the plaque, and plaque volume; and Optical Coherence Tomography (OCT) allows physicians to assess tears in the surface of plaque and plaque thickness; to evaluate high risk non-infarct-related coronary lesion in patients who have suffered a recent heart attack, underwent successful opening of the artery with a stent, and have blockages greater than or equal to 50% in one or more of the other arteries to the heart; and to correlate this findings with cardiovascular outcomes at 1 year.

DETAILED DESCRIPTION:
This is a prospective, open-label, single center registry. The study is designed to characterize plaque (i.e., assess vulnerable plaque features such as plaque tears, plaque thickness, plaque volume, and lipid content in plaque) in heart arteries in patients who have suffered a recent acute heart attack, and who have blockages >50% in one or more of the other arteries in the heart. The procedure to do this will not be the same procedure that was done to open the artery that caused the heart attack, but will be scheduled 2-40 days after the first procedure, depending on the urgency to evaluate the other arteries and the stability of the patient after the first procedure. The study will specifically evaluate the plaque characteristics in the arteries that didn't cause the heart attack, to see if these arteries have vulnerable plaque and is at risk for future heart attacks. If FFR shows abnormal blood flow, these arteries will be treated with stents. All patients will be followed for 12 months after the second catheterization. The purpose of the study is to determine how commonly vulnerable plaques are identified in patients with acute heart attacks, and how often these lead to future cardiac problems. Identification of plaque features that lead to future problems may allow the development of new medications and devices to prevent future heart attacks and death. These same plaque features are also thought to be operative in patients with blockages in the arteries to the brain, so this study may have important implications for stroke prevention as well. All patients will be considered eligible for participation if they had a recent acute heart attack resulting from complete occlusion of an artery to the heart, if the stent procedure to open the artery was successful, and if they have blockages > 50% in at least one other major heart artery. Patients will not be eligible for participation if they are too unstable with regard to heart, lung, brain, or kidney function, or if they have previous bypasses to the heart.

In selected patients, Coronary CT Angiography (CCTA) will be performed after the initial procedure to open the artery within 40 days. CCTA images will be evaluated for plaque characteristics, and correlated with the invasive findings.Fractional flow reserve via computed tomography (FFRCT), a non-invasive computed tomography method of measuring blood flow in the blocked arteries; will also be determined and correlated with invasive FFR.

The standard portion of the procedure includes the angiogram (X-ray pictures of the arteries), FFR (measurement of blood flow in the artery), IVUS and/or OCT (to assess the diameter of the artery and the size of the stent), medications, and all office visits. The research portion of the study requires all imaging studies be performed (NIRS IVUS, OCT, FFR) rather than just one or two of these imaging studies, and the CCTA.

ELIGIBILITY:
Inclusion Criteria:

All patients with ST-elevation acute myocardial infarction (STEMI) and age > 18 years who meet all of the following criteria:

* Successful primary Percutaneous Intervention (PCI) of the Infarcted Related Artery (IRA) defined as final stenosis < 30%, Thrombolysis In Myocardial Infarction (TIMI) 3 flow
* At least 1 non-IRA with diameter stenosis ≥ 50% and reference vessel diameter > 2mm
* None of the exclusion criteria

Exclusion Criteria:

Patients will be excluded if any of the following are present:

* Cardiogenic shock that persists > 24 hours after primary PCI
* Diffuse disease in non-IRA that precludes successful stenting
* Estimated Glomerular Filtration Rate (eGFR) < 30 cc/min/1.73 m2 after hydration or optimization of Congestive Heart Failure (CHF) for cardiac death
* eGFR <60 cc/min/1.73 m2, will be in the MIAMI study for invasive imaging treatment group/cohort but will not get the coronary CCTA
* eGFR < 60 cc/min/1.73 m2, for coronary CCTA
* Active bleeding as defined as a fall in hemoglobin (HGB) concentration > 3 g/dL within 24 hours requiring blood transfusion, vasopressors to maintain Systolic BP > 100mmhg, or emergency surgical, endovascular, or endoscopic intervention.
* Mechanical complication of MI such as severe Mitral-Valve Regurgitation (MR), Ventricular Septal Defect (VSD) or pulmonary edema
* Uncontrolled Ventricular Tachycardia (VT) after primary PCI
* Inability to provide informed consent
* Ventilator-dependent respiratory failure
* Only non-IRA is a chronic total occlusion
* Non-IRA is in a Saphenous Vein Graft (SVG) or arterial graft
* Non-IRA is in the left main, ostial Left Anterior Descending (LAD), or ostial Left circumflex (LCX)
* Non-IRA includes a bifurcation with side branch > 2mm, medina 1-1-1
* Need for multivessel primary PCI during the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of hemodynamically-significant stenosis and "vulnerable" plaque in non-infarct-related coronary arteries in STEMI patients as measured during cardiac cath | 40 Days
  2-40 days after the first cardiac catheterization procedure, depending on the urgency to evaluate the other arteries and the stability of the patient after the first procedure. Repeat cardiac catheterization for Data Analysis Stenosis severity (using angiographic criteria defined as Diameter Stenosis (DS) > 70% and DS > 50%;
Prevalence of hemodynamically-significant stenosis and "vulnerable" plaque in non-infarct-related coronary arteries in STEMI patients as measured by IVUS | 40 Days
  Stenosis severity will be measured by IVUS criteria defined as minimal lumen cross sectional area (mCSA) < 4mm2, mCSA < 2.5mm2, plaque volume; and vulnerable plaque by IVUS-fibrous cap thickness.
Prevalence of hemodynamically-significant stenosis and "vulnerable" plaque in non-infarct-related coronary arteries in STEMI patients as measured by FFR | 40 Days
  cardiac catheterization with FFR criteria defined as FFR < 0.80;
Prevalence of hemodynamically-significant stenosis and "vulnerable" plaque in non-infarct-related coronary arteries in STEMI patients as measured by OCT | 2 - 40 Days
  Vulnerable plaque characteristics will be measured by OCT criteria - plaque ulceration, erosion, thrombus, fibrous cap thickness
Prevalence of hemodynamically-significant stenosis in non-infarct-related coronary arteries in STEMI patients as measured by CCTA | 2 - 40 Days
  Stenosis severity will be measured by CCTA criteria-Diameter Stenosis >70%
Prevalence of hemodynamically-significant stenosis and "vulnerable" plaque in non-infarct-related coronary arteries in STEMI patients as measured by NIRS | 2 - 40 Days
  Vulnerable plaque characteristics will be measure by NIRS criteria - Lipid Core Burden Index (LCBI) - 4mm > 300, Lipid Core Containing Plaque (LCP) distribution

SECONDARY OUTCOMES:
Incidence of cardiac events at 1-year after STEMI. | 1 Year
  Correlation between cardiovascular outcomes (MACE) at 1-year with measures of stenosis severity and presence of ≥ 1 feature of vulnerable plaque.
Correlation with coronary angiography with imagings findings and Coronary CT Angiography (CCTA) imaging findings. | 40 Days
  In selected patients, Coronary CT Angiography (CCTA) will be performed within 40 days after the initial procedure that opens the artery . CCTA images will be evaluated for plaque characteristics, and correlated with the invasive findings.Fractional flow reserve via computed tomography (FFRCT), a non-invasive computed tomography method of measuring blood flow in the blocked arteries; will also be determined and correlated with invasive FFR.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Safian, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beamont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ihdayhid AR, Tzimas G, Peterson K, Ng N, Mirza S, Maehara A, Safian RD. Diagnostic Performance of AI-enabled Plaque Quantification from Coronary CT Angiography Compared with Intravascular Ultrasound. Radiol Cardiothorac Imaging. 2024 Dec;6(6):e230312. doi: 10.1148/ryct.230312. PMID 39540820